CLINICAL TRIAL: NCT06215742
Title: A Randomized Controlled Study to Explore Clinical Effect of Stellate Ganglion Block on Gastroesophageal Reflux Disease
Brief Title: Clinical Effect of Stellate Ganglion Block on Gastroesophageal Reflux Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: ethical issues
Sponsor: Zeng Changhao (Other)
Responsible Party: Sponsor-Investigator, Zeng Changhao, Research Director, People's Hospital of Zhengzhou University
Organization: People's Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-KY-0110
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the experimental group (Experimental): The study lasts 20d for each patient. During the treatment, All the participants are provided with the rehabilitation therapy. Based on this, the patients in the experimental group are provided with Stellate Ganglion Block , using 1.5ml of 2% Lidocaine hydrochloride (1ml: 0.5mg) and 500ug of Vitamin B12 (1ml: 0.5g), once a day.
  Interventions: Behavioral: Rehabilitation therapy; Procedure: Stellate ganglion block
- the control group (Active Comparator): The study lasts 20d for each patient. During the treatment, All the participants are provided with the rehabilitation therapy.
  Interventions: Behavioral: Rehabilitation therapy

INTERVENTIONS:
Behavioral: Rehabilitation therapy — Rehabilitation therapy includes
  1. Diet management: Avoiding consumption of irritant foods and beverages, such as spicy foods, caffeine, alcohol, and acidic foods. Controlling portion sizes and meal timing, and adopting smaller, more frequent meals.
  2. Lifestyle adjustments: Avoiding lying down or bending immediately after meals, maintaining a sitting or upright position for at least 2 hours. Adjusting sleeping positions by elevating the head of the bed to reduce nighttime acid reflux. Avoiding excessive exertion and managing stress levels.
  3. Rehabilitation training: Strengthening the control of esophageal and gastric muscles through rehabilitation exercises to improve the function of the gastroesophageal sphincter and prevent gastric fluid reflux.
Procedure: Stellate ganglion block — Based on the invention above, the patients in the observation group were provided with Stellate ganglion block, using 1.5ml of 2% Lidocaine hydrochloride (1ml: 0.5mg) and 500ug of Vitamin B12 (1ml: 0.5g). The percutaneous approach via the paratracheal route was used for Stellate ganglion block. The operator stood on the side of the block, instructed the patient to lie supine with a thin pillow placed below the shoulders, and tilted the head 45° towards the blocked side, fully exposing the neck. Then, routine disinfection of the neck skin was performed. The puncture site was located 2.5 cm above the sternoclavicular joint and 1.5 cm lateral to the midline of the neck.
  Arms: the experimental group

SUMMARY:
The goal of this clinical trial is to explore Clinical Effect of Stellate Ganglion Block on Gastroesophageal Reflux Disease. The main question it aims to answer is:

• Can stellate ganglion block improve gastroesophageal reflux symptoms better on the basis of rehabilitation training? Participants will be randomly allocated into the control group or the experimental group, all under rehabilitation treatment, the experimental group will be given Stellate Ganglion Block once a day additionally. The study lasts 20 days for each participant. Researchers will compare the Gastroesophageal Reflux Disease Questionnaire, Pressure pain threshold, Self-Evaluation Questionnaire for Gastroesophageal Reflux Disease, to see if the Stellate Ganglion Block can help improve the symptom.

DETAILED DESCRIPTION:
Gastroesophageal reflux is a common digestive disorder characterized by the backflow of stomach contents and fluids into the esophagus.

The goal of this clinical trial is to explore Clinical Effect of Stellate Ganglion Block on Gastroesophageal Reflux Disease. The main question it aims to answer is:

• Can stellate ganglion block improve gastroesophageal reflux symptoms better on the basis of rehabilitation training? Participants will be randomly allocated into the control group or the experimental group, all under rehabilitation treatment, the experimental group will be given Stellate Ganglion Block once a day additionally. The study lasts 20 days for each participant. Researchers will compare the Gastroesophageal Reflux Disease Questionnaire, Pressure pain threshold, Self-Evaluation Questionnaire for Gastroesophageal Reflux Disease, to see if the Stellate Ganglion Block can help improve the symptom.

ELIGIBILITY:
Inclusion Criteria:

* Gastroesophageal Reflux Disease diagnosis after determination of acid reflux by gastroenterologist, with upper endoscopy and/or impedance-pHmetry, which confirmed esophagitis and/or hiatal hernia.
* aged between 18 and 80 years old.
* subjects who tolerate cervical movements in sitting position.
* stable vital signs.
* normal consciousness

Exclusion Criteria:

* contraindications for stellate ganglion block.
* peptic ulcer.
* previous or present gastric cancer.
* previous gastric surgery.
* recent fractures or cervical trauma.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
Gastroesophageal Reflux Disease Questionnaire | day 1 and day 20
  The Gastroesophageal Reflux Disease Questionnaire is a commonly used questionnaire for assessing the symptoms and severity of gastroesophageal reflux disease. It was developed by gastrointestinal experts in Germany and consists of six questions that evaluate the frequency and severity of gastroesophageal reflux disease symptoms. For each question, patients are required to select the answer that best corresponds to their situation. Different scores are assigned based on the chosen answers, and a total score is calculated at the end.
  The maximum score for the Test is 12 points, with a lower score indicating milder symptoms and a higher score indicating more severe symptoms.

SECONDARY OUTCOMES:
Pressure pain threshold | day 1 and day 20
  Pressure is applied on the spinous processes of the fourth cervical vertebrae. Pressure will be uniformly increased, and patients are given the identical instruction, "let me know when the sensation of pressure becomes uncomfortable or painful". At this point, the pressure will be immediately released, and the plunger is retracted by the evaluator. And the pressure will be recorded
Modified Mayo Clinic Dysphagia-30 questionnaire | day 1 and day 20
  Modified Mayo Clinic Dysphagia-30 questionnaire is a standardized tool used to assess the severity and impact of dysphagia on patients' daily lives. The questionnaire consists of 30 items that evaluate several aspects of swallowing function, including swallowing ability, eating habits, and quality of life. The total score for the Modified Mayo Clinic Dysphagia-30 questionnaire is 120 points, and a lower score indicates milder symptoms and less impact on daily life.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Study Director — Site Coordinator of United Medical Group located in Miami
Locations (1):
- Zheng Da yi Yuan Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No